CLINICAL TRIAL: NCT05114707
Title: Camrelizumab Plus Chemoradiotherapy for Patients With Locoregional Cancer of Nasal Cavity and Paranasal Sinuses: a Phase II Multicenter Study
Brief Title: Camrelizumab Plus Chemoradiotherapy for Patients With Locoregional Cancer of Nasal Cavity and Paranasal Sinuses
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Fei Han, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2021-040-01
Record Dates: First submitted 2021-10-31; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Nasal Cavity Cancer; Paranasal Sinus Cancer; Camrelizumab; Induction Chemotherapy; Intensity Modulated Radiotherapy; Concurrent Chemotherapy
MeSH Terms: conditions — Paranasal Sinus Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- camrelizumab group (Experimental)
  Interventions: Drug: camrelizumab

INTERVENTIONS:
Drug: camrelizumab — Camrelizumab was administrated with 200mg each time, every three weeks for a total of 11 cycles since the first day of induction chemotherapy.

SUMMARY:
Patients with locoregional cancer of nasal cavity and paranasal sinuses are candidate for this study. All the eligible patients receive three cycles of induction chemotherapy (docetaxel 60mg/m2+cisplatin 60mg/m2+5-FU2.5g/m2,civ48h, q3w) followed by concurrent two cycles of cisplatin (80mg/m2,q3w) with curative intensity modulated radiotherapy. Besides, camrelizumab (200mg) is administrated every three weeks for a total of 11 cycles since the first day of induction chemotherapy. We aim to evaluate the three years failure free survival of these patients by the combination of camrelizumab with curative radiotherapy and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed squamous cancer of nasal cavity and paranasal sinuses
* T4bN0-3M0 (AJCC8th) or unresectable lymph nodes or refusal of surgery
* KPS≥70
* NE≥ 1.5×10E9/L, HGB ≥ 100g/L and PLT ≥100×10E9/L
* ALT≤ 1.5 upper limit of normal (ULN), AST≤ 1.5ULN and bilirubin ≤ 1.5ULN
* creatinine clearance rate ≥ 60 ml/min (calculated by Cockcroft-Gault)

Exclusion Criteria:

* older than 65 or younger than 18
* HBsAg (+) and HBV DNA >1×10E3 copiers /mL
* HCV (+)
* HIV (+)
* autoimmune diseases
* interstitial lung diseases
* had other cancers before

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2024-04-16 (Estimated); Study Completion 2024-04-16 (Estimated)

PRIMARY OUTCOMES:
3-year failure free survival | 3-year
  time from the randomization to the first treatment failure or death

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No